CLINICAL TRIAL: NCT00510549
Title: A Prospective, Randomized, Multicenter, Open Label, Interventional Pilot Study To Compare Mortality, Morbidity and QOL in Hemodialysis Versus Peritoneal Dialysis Subjects
Brief Title: Comparison of the Impact of Dialysis Treatment Type on Patient Survival
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Baxter Healthcare Corporation, Company
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SurvivalHD/PDFinal 28/03/2007
Record Dates: First submitted 2007-07-16; First posted 2007-08-02 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, PD (Active Comparator): Peritoneal Dialysis
  Interventions: Procedure: Modality: Peritoneal Dialysis
- 2, HD (Active Comparator): Hemodialysis
  Interventions: Procedure: Modality: Peritoneal Dialysis

INTERVENTIONS:
Procedure: Modality: Peritoneal Dialysis — Peritoneal Dialysis: CAPD; Hemodialysis: 3 times/week

SUMMARY:
As the influence of type of dialysis on survival of end stage renal disease (ESRD) patients remains unanswered, the present study is designed (randomized, prospective, multicenter, interventional) to assess clinical outcomes, and compare mortality, morbidity, Quality of Life (QOL) and cost effectiveness between maintenance In-center Hemodialysis (ICHD) and Continuous Ambulatory Peritoneal dialysis (CAPD). These data will ultimately bring clarity on whether or not any difference in patient survival exists between the two modalities.

In order to test the feasibility of patients' willingness to be randomized to two different modality groups and retained in the randomized group, a pilot study is planned before the conduct of a main study.

This pilot study comprises of a 6 months study, plus a 6 months observation if there is possibility to switch the patients into the main study.

All ESRD patients requiring dialysis treatment within 8 weeks after a pre-study visit will be recorded in each site. Patients who provide written inform consent for collecting relevant information will be screened using certain inclusion/exclusion criteria. Eligible patients will undergo a standardized education regarding ESRD and treatment options. Thereafter the patient will be required to provide a second inform consent allowing for randomization and entrance into the study. Eligible patient will be randomized to either PD or HD treatment.

The patients will be followed for a period of 6 months, during which patients will be treated with PD or HD as prescribed at each site, while meeting the dialysis adequacy and other indicators. For the first 3 months monthly visits are required, after which an every 3 months visit is planned.

In this pilot study, the main objective is to assess the willingness of ESRD patients to be randomized to either PD or HD treatment; thereby determining if an adequate number of eligible patients can be recruited for a future large-scale study.

DETAILED DESCRIPTION:
refer to brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are at least 18 years of age.
2. Patients who have read, understood and given written informed consent after the nature of the study has been explained.
3. Patients who have a diagnosis of ESRD (GFR ≤ 10 ml/min), without a permanent access for dialysis.
4. Patients who are able to comprehend a modality education program.
5. Patients who are judged as capable of being trained for home based PD.
6. Patients as justified by their physicians requiring dialysis treatment within 6 weeks after randomization (Patients who require urgent temporary dialysis before randomization may also be eligible for recruitment after being stabilized with temporary HD or PD)
7. Patients who are expected to remain on dialysis for at least 6 months.
8. Patients must have a negative HIV test at screening. -

Exclusion Criteria:

1. Patients that have already received a permanent catheter or access that is intended for permanent therapy use before receiving modality information, or have already received permanent dialysis (If an access is present within 4 weeks prior to screening for back-up purposes, or for acute treatment for life threatening uremic symptoms, electrolyte abnormalities or fluid overload, this does not exclude the patient from enrollment).
2. Patients who previously have received renal transplantation and are still prescribed immunosuppressive therapy.
3. Patients who are unwilling or unable to follow the protocol.
4. Patients with concomitant participation in any other interventional study, or who have received any investigational drug, biologic or device within five half-lives of the physiological action or 30 days, whichever is longer, prior to screening.
5. Patients justified as not eligible for either PD or HD due to:

   * PD: documented extensive intra-peritoneal adhesions, severe infective skin disorder, or other situation contradicting PD (eg., active inflammatory bowel disease)
   * HD: severe cardiac instability and inability to a gain permanent vascular access.
6. Patients who have a history of drug or alcohol abuse within the six months prior to entering the study
7. Patients who have active systemic infections, such as tuberculosis, septicemia or systemic fungal infections.
8. Patients who have malignancies requiring active chemotherapy or radiation therapy.
9. The presence of other terminal illness likely to cause death within 6 months
10. Patients who have any other serious acute or active conditions that in the investigator's opinion would preclude their participation in the study.
11. Female patients who are pregnant, lactating or planning on becoming pregnant during the study period.
12. Patients who are allergic to starch-based polymers, maltose or isomaltose
13. Patients who have glycogen storage disease.
14. Patients who have a significant psychiatric disorder or mental disability that could interfere with the patient's ability to provide informed consent and/or comply with protocol procedures -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess willingness of ESRD patients to be randomized to either PD or HD; thereby determining if an adequate number of eligible patients can be recruited for a future large-scale study. | August 2008

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Qi QIAN, Prof, Principal Investigator — Center for one Baxter -Tel: 8004229837; Tao Wang, Prof, Principal Investigator — Center for one Baxter -Tel: 8004229837
Locations (2):
- China (2):
  - Bejing No.3 Hospital, Beijing
  - Renji Hospital, Shanghai, Shanghai

REFERENCES:
- [Derived] Ethier I, Hayat A, Pei J, Hawley CM, Johnson DW, Francis RS, Wong G, Craig JC, Viecelli AK, Htay H, Ng S, Leibowitz S, Cho Y. Peritoneal dialysis versus haemodialysis for people commencing dialysis. Cochrane Database Syst Rev. 2024 Jun 20;6(6):CD013800. doi: 10.1002/14651858.CD013800.pub2. PMID 38899545